CLINICAL TRIAL: NCT05785715
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Dose, Multicenter Phase 2 Induction Study With Long-Term Extension to Evaluate the Clinical Activity and Safety of Oral NX-13 in Participants w/ Moderate to Severe Ulcerative Colitis
Brief Title: Study to Evaluate the Clinical Activity and Safety of Oral NX-13 in Moderate to Severe Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision_Not Safety Related
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NX-13-201
Record Dates: First submitted 2023-02-13; First posted 2023-03-27 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; moderate; severe
MeSH Terms: conditions — Colitis, Ulcerative; Lymphoma, Follicular | interventions — NX-13

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NX-13 250mg (Experimental): Subjects will take study drug by ingesting three tablets per day, recommended at the same time daily for consistency. Subjects in a NX-13 group will receive either 250 mg or 750 mg of NX-13 in 3 tablets and subjects in the placebo group will receive matching placebo.
  Interventions: Drug: NX-13 250mg
- NX-13 750mg (Experimental): Subjects will take study drug by ingesting three tablets per day, recommended at the same time daily for consistency. Subjects in a NX-13 group will receive either 250 mg or 750 mg of NX-13 in 3 tablets and subjects in the placebo group will receive matching placebo.
  Interventions: Drug: NX-13 750mg
- NX-13 Placebo (Placebo Comparator): Subjects will take study drug by ingesting three tablets per day, recommended at the same time daily for consistency. Subjects in a NX-13 group will receive either 250 mg or 750 mg of NX-13 in 3 tablets and subjects in the placebo group will receive matching placebo.
  Interventions: Drug: NX-13 Placebo

INTERVENTIONS:
Drug: NX-13 250mg — NX-13 250mg tablet, plus 2 placebo tablets
  Arms: NX-13 250mg
Drug: NX-13 750mg — NX-13 250mg tablets times 3 to equal 750mg
  Arms: NX-13 750mg
Drug: NX-13 Placebo — NX-13 Placebo tablets times 3 for blinding purposes
  Arms: NX-13 Placebo

SUMMARY:
Phase 2 induction study with a long-term extension (LTE) period in participants with moderate to severe ulcerative colitis (UC).

DETAILED DESCRIPTION:
This is a randomized, multicenter, double-blind, placebo-controlled, multiple dose exploratory Phase 2 induction study with a long-term extension (LTE) period in participants with moderate to severe ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects aged 18 to 75 years (inclusive)
* Diagnosis of UC ≥ 90 days before screening confirmed by histologic evidence
* Active UC defined as a total Mayo Score (MMS) of ≥ 5 (inclusive) at baseline
* ES ≥ 2 within 14 days prior to randomization
* RBS ≥ 1.

Exclusion Criteria:

* Severe extensive colitis as evidenced by physician judgment that the participant is likely to require hospitalization for medical care or surgical intervention of any kind for UC (e.g., colectomy) within the 12 weeks after randomization;
* Current evidence of fulminant colitis, toxic megacolon or recent history (within 6 months prior to screening) of toxic megacolon, or bowel perforation
* Diagnosis of Crohn's disease (CD) or indeterminate colitis, or the presence or history of a fistula consistent with CD
* Diagnosis of microscopic colitis, ischemic colitis, or radiation colitis
* Bacterial or parasitic pathogenic enteric infection;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
To assess the clinical activity of oral NX-13 vs placebo | 365 days
  Change from baseline in mean Modified Mayo Score (MMS) vs placebo. Total score Modified Mayo score 0-9, with higher scores representing more severe disease activity.

SECONDARY OUTCOMES:
Safety and Tolerability-AE/SAE - Hematology | 365 days
  Treatment Emergent Adverse Event/Serious Adverse Event (TEAEs/SAEs) related to hematology. Assessment will be made by summarizing the percentage of subjects with changes from baseline through routine hematology panel (white blood cells, red blood cells, Hemoglobin, Hematocrit, and platelets). All biomarkers are exploratory objectives.
Safety and Tolerability-AE/SAE - Chemistry | 365 days
  Treatment Emergent Adverse Event/Serious Adverse Event (TEAEs/SAEs) related to chemistry. Assessment will be made by summarizing the percentage of subjects with changes from baseline through routine chemistry panel (Blood Urea Nitrogren creatinine, Creatine Kinase bilirubin, Aspartate aminotransferase (AST), Alanine transaminase (ALT), Alkaline phosphatase (ALP), Sodium (Na), Potassium (K), Chloride (CL), bicarb, Calcium (CA), Magnesium (MG), Phosphorus, uric acid, total protein, albumin, glucose, Gamma-glutamyl transferase (GGT), total cholesterol, Low-density lipoprotein (LDL), High-density lipoprotein (HDL), and triglycerides) urinalysis, Estimated Glomerular filtration rate (eGFR). All biomarkers are exploratory objectives.
Safety and Tolerability-AE/SAE - Vital Signs | 365 days
  Treatment Emergent Adverse Event/Serious Adverse Event (TEAEs/SAEs) related to vital signs. Assessment will be made by summarizing the percentage of subjects with changes from baseline through (sitting blood pressure, resting heart rate, and temperature). Changes from baseline deemed clinically significant or associates with AEs (heart rate, pulse rate, QRS, QT, and correct QT).

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie, Study Director — AbbVie
Locations (35):
- United States (11):
  - Miami Clinical Research, Miami, Florida
  - Orlando Health, Inc., Orlando, Florida
  - GCP Clinical Research, Tampa, Florida
  - Digestive Health Center of Michigan, Chesterfield, Michigan
  - Clinical Research Institute of Michigan, Troy, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Digestive Disease Specialist, Inc-INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Digestive Health Associates of Texas-GI Alliance Research-Garland, Garland, Texas
  - Digestive Health Associates of Texas-GI Alliance, Mansfield, Texas
  - Texas Digestive Disease Consultants-GI Alliance Research, Southlake, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven, Belgium
- Italy (5):
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera - Universitaria Sant' Andrea, Roma
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Istituto Clinico Humanitas, Rozzano
  - IRCCS Fondazione Casa Sollievo della Sofferenza SG Rotondo, San Giovanni Rotondo
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
- Poland (18):
  - ClinSante - Ośrodek Badań Klinicznych w Bydgoszczy, Bydgoszcz
  - Przychodnia Vitamed NFZ, Bydgoszcz
  - AmiCare Centrum Medyczne, Jelenia Góra
  - VITA LONGA Clinic - Katowice, Katowice
  - Krakowska Przychodnia FutureMeds, Krakow
  - AmiCare Sp. z o.o. Sp.k., Lodz
  - Amicare Sp z o.o. S.K, Opoczno
  - Twoja Przychodnia Opolskie Centrum Medyczne, Opole
  - RiverMED Poradnie Specjalistyczne Poznań, Poznan
  - Endoskopia Sp. z o.o., Sopot
  - Sonomed Sp. z o.o. Centrum Medyczne, Szczecin
  - Twoja Przychodnia Szczecińskie Centrum Medyczne, Szczecin
  - Torunskiego Centrum Gastrologii I Endoskopii - Gastromed, Torun
  - H-T Centrum Medyczne, Tychy
  - Office of Jaroslaw Kierkus, Dr N Med, Warsaw
  - Centrum Badań Klinicznych Piotr Napora Lekarze Sp. p., Wroclaw
  - Zabobrze Centrum Medyczne, Wroclaw
  - Centrum Diagnostyczno - Lecznicze Barska, Włocławek

IPD SHARING:
Plan to Share IPD: No